CLINICAL TRIAL: NCT04115826
Title: Per-oral Pancreatoscopy-guided Lithotripsy vs. Extracorporeal Shock Wave Lithotripsy in Chronic Pancreatitis
Brief Title: ESWL vs. Pancreatoscopy-guided Lithotripsy for Painful Chronic Calcific Pancreatitis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-0402
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Pancreatitis, Chronic
Keywords: pancreatic duct stone; extracorporeal shock-wave lithotripsy; pancreatoscopy; quality of life; chronic pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Lithotripsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigator interpreting final stone clearance pancreatograms will be blinded to the intervention received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal Shock-Wave Lithotripsy (Placebo Comparator): Stone localization will first be performed by obtaining high-quality plain films of the pancreatic area in left and right oblique positions using a two-dimensional radiologic targeting system.Depending on the stone localization, ESWL will then be performed with the patient in either slight left or right lateral decubitus with shock waves entering the body from the ventral side. The shockwaves will be focused first on the most distally located stone within the main duct and then on other calculi moving from the head towards the body. If a stent has been inserted during preceding ERP then this may also serve as a guide to target main pancreatic duct stones by ESWL. A total of one hour of ESWL at a rate of 60-120 shocks/minute will be delivered in one treatment session.
  Interventions: Procedure: Extracorporeal Shock-Wave Lithotripsy
- Per-oral Pancreatoscopy-guided Lithotripsy (Active Comparator): Standard ERP will be performed to cannulate the PD, perform pancreatic sphincterotomy, and stricture dilation as necessary. A pancreatoscope (Spyglass Digital System, Boston Scientific, Marlborough, MA) will then be inserted through the duodenoscope into the PD. For PPL, electrical pulses will be delivered through an aqueous medium by EHL or LL with the probe tip in contact with or 1-2mm away from the stone. Settings for EHL (1.9F fiber; Autolith, Northgate Technologies, Elgin, IL) are 10-20 pulses/second with a power of 50-100; and for LL (200, 272, or 365 micrometer fiber, Versa Pulse Power Suite 20-W Holmium laser, New Star, Roseville, CA) ranging from 0.8 - 2.5 Joules with a frequency of 8-15Hz and power of 9-30 W. A maximum of 1 hour of intraductal lithotripsy will be allowed to reduce performance bias.
  Interventions: Procedure: Per-oral Pancreatoscopy-guided Lithotripsy

INTERVENTIONS:
Procedure: Per-oral Pancreatoscopy-guided Lithotripsy — Per-oral Pancreatoscopy-guided lithotripsy will be administered for a maximum of 4 sessions (1 hour max per session). Either electrohydraulic lithotripsy or laser lithotripsy will be allowed during the session at the discretion of the endoscopist.
  Arms: Per-oral Pancreatoscopy-guided Lithotripsy
Procedure: Extracorporeal Shock-Wave Lithotripsy — ESWL will then be performed with the patient in either slight left or right lateral decubitus with shock waves entering the body from the ventral side. The shockwaves will be focused first on the most distally located stone within the main duct and then on other calculi moving from the head towards the body. If a stent has been inserted during preceding ERP then this may also serve as a guide to target main pancreatic duct stones by ESWL. A total of one hour of ESWL at a rate of 60-120 shocks/minute will be delivered in one treatment session.
  Arms: Extracorporeal Shock-Wave Lithotripsy

SUMMARY:
This is a multi-center randomized controlled trial comparing extracorporeal shock-wave lithotripsy (ESWL) with per-oral pancreatoscopy-guided lithotripsy (PPL) in the treatment of patients with chronic pancreatitis and refractory main pancreatic duct stones. This study will be comparing the two treatment options for patients who have stones that fail initial endoscopic therapy via endoscopic retrograde pancreatography (ERCP). The study will look at the stone clearance rates and patient-centered outcomes including quality of life and pain.

DETAILED DESCRIPTION:
Patients with chronic pancreatitis frequently develop obstructing pancreatic duct stones which can lead to severe pain. Current standard methods to remove these stones include ERCP and extracorporeal shock-wave lithotripsy (ESWL) which are limited in removing larger and multiple impacted stones. Availability in the USA of ESWL for this indication also may be limited even at major referral centers. The introduction of single-operator per-oral pancreatoscopy (SpyGlassTM) has enabled direct intraductal visualization to target stones. Retrospective studies demonstrate a high success rate but literature is quite limited, uncontrolled, and highly selective. Further, many experts and recent European Society Guidelines suggest that ESWL is the only primary therapy for larger stones (5mm or larger) and that intraductal endoscopy and lithotripsy should only be used for 'salvage' therapy in select patients.

A critical need exists to compare the efficacy of per oral pancreatoscopy-guided lithotripsy (PPL) with ESWL to determine which therapy is most efficacious in removing refractory PD stones. The investigators believe ERCP with POP has distinct advantages of localizing 'shocks' to the stones, helping to identify and treat underlying strictures in the duct, and lithotripsy of multiple stones can be performed at a single session with a recent multi-center international retrospective study showing all stones removed in a single session in over 70% of cases. Therefore, this project seeks to change the perceived standard of care as it relates to symptomatic pancreatic duct stones in this population, shifting the pendulum towards endoscopic and specifically pancreatoscopy-guided therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18-89
2. Subjects with abdominal pain secondary to chronic calcific pancreatitis and main pancreatic duct stones found on cross-sectional imaging, EUS, or ERP with upstream PD dilation
3. Main PD stones in the head or body that are greater than 50% in size of the immediate downstream diameter of the pancreatic duct
4. Stones ≥ 5 mm in diameter or impacted in the main PD on cross-sectional imaging or EUS

Exclusion Criteria:

1. Subjects who have previously received PPL or ESWL for PD stones within 12 months of enrollment
2. Patients with PD stones isolated in the tail or side branches of the main duct
3. Pancreatic tail stones comprising more than one-third of the stone burden within the main PD, if multiple locations of stones are noted within the main PD
4. Nontraversable ansa loop with upstream stones
5. Inability to place a transpapillary pancreatic duct stent during ERP
6. Patients with prior pancreatic surgery or surgically altered gastroduodenal anatomy, such as Roux-en-Y surgery
7. Acquired pancreas divisum
8. Significant cardiopulmonary co-morbidities precluding general anesthesia
9. Patients with coagulation disorders that cannot be corrected to an INR below 2.0
10. Patients with ongoing alcohol abuse and/or illicit drug use, except products containing THC
11. Pregnancy
12. Patients in active treatment for malignancy other than non-melanoma skin cancer or papillary thyroid cancer

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Stone Clearance Rate | Up to 4 hours (four 1-hour sessions)
  The rate of complete clearance of the main pancreatic duct of all stones.

SECONDARY OUTCOMES:
Change In Quality of Life as Measured Using PANQOLI Score | At the conclusion of treatment success/failure at 1,3,6, and 12 months follow-up
  Change in quality of life as measured using the PANQOLI (PANcreatitis Quality of Life Instrument), a chronic pancreatitis-specific quality of life instrument. This instrument has a score range from 0 to 100, which higher scores denoting better quality of life. The questionnaire has 18 items and questions 1, 2, 3, 4, 5, 6, 12, 13, 14, 15, 16, 17, and 18 are reverse scored while items 7, 8, 9, 10, and 11 are scored at face value. The final score is the sum of the scores from all 18 questions.
Change in Pain Levels as Measured Using the COMPAT Score | At the conclusion of treatment success/failure at 1,3,6, and 12 months follow-up
  Change in pain levels as measured using the comprehensive pain assessment tool, (COMPAT), a chronic pancreatitis-specific pain questionnaire. The questionnaire consists of 23 questions. A score is assessed for question # 14, which consists of 28 questions with scores ranging from 0 to 10, with 10 representing worse pain. A maximum score of 280 is possible for this component of the COMPAT.

CONTACTS AND LOCATIONS:
Overall Officials: Raj J Shah, MD, Principal Investigator — University of Colorado Anschutz Medical Campus, Professor of Medicine
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available to researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available at the conclusion of the study once the results are published.
Access Criteria: Formal proposal required

REFERENCES:
- [Derived] Han S, Miley A, Akshintala V, Freeman ML, Kahaleh M, Othman M, Patel S, Papachristou GI, Raijman I, Sankey N, Sayana H, Singh V, Tarnasky P, Trikudanathan G, Shah RJ. Per-oral pancreatoscopy-guided lithotripsy vs. extracorporeal shock wave lithotripsy for treating refractory main pancreatic duct stones in chronic pancreatitis: Protocol for an open-label multi-center randomized clinical trial. Pancreatology. 2022 Dec;22(8):1120-1125. doi: 10.1016/j.pan.2022.09.245. Epub 2022 Oct 15. PMID 36273991

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: POP x ESWL Protocol (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT04115826/Prot_SAP_ICF_002.pdf
  • Informed Consent Form: POP x ESWL ICF (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT04115826/ICF_003.pdf